CLINICAL TRIAL: NCT05689177
Title: Humoral Immunity Study After a Booster Dose of Soberana Plus (FINLAY-FR-1A) Vaccine Against COVID-19 (Republic of Cuba)
Brief Title: Humoral Immunity Study After a Booster Dose of Soberana Plus (FINLAY-FR-1A) Vaccine Against COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Gomel State Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GomelSMU
Record Dates: First submitted 2023-01-16; First posted 2023-01-19 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Humoral Immunity
Keywords: COVID-19; SARS-CoV-2; Humoral immunity; Booster dose
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Booster dose administration to younger participants (Experimental): Participants 18-25 y.o. take a booster dose of vaccine against COVID-19 (Soberana Plus (FINLAY-FR-1A), Republic of Cuba)
  Interventions: Biological: Protein subunit vaccine Soberana Plus (FINLAY-FR-1A) is a vaccine against COVID-19 produced by The Finlay Vaccine Institute and The Centre of Molecular Immunology (Republic of Cuba)
- Booster dose administration to older participants (Experimental): Participants 26-80 y.o. take a booster dose of vaccine against COVID-19 (Soberana Plus (FINLAY-FR-1A) Republic of Cuba)
  Interventions: Biological: Protein subunit vaccine Soberana Plus (FINLAY-FR-1A) is a vaccine against COVID-19 produced by The Finlay Vaccine Institute and The Centre of Molecular Immunology (Republic of Cuba)

INTERVENTIONS:
Biological: Protein subunit vaccine Soberana Plus (FINLAY-FR-1A) is a vaccine against COVID-19 produced by The Finlay Vaccine Institute and The Centre of Molecular Immunology (Republic of Cuba) — Booster dose administration

SUMMARY:
To evaluate the dynamics of IgG levels to the SARS-CoV-2 virus after a booster dose of Soberana Plus vaccine.

DETAILED DESCRIPTION:
Prospective clinical study of evaluation of the immune response to booster dose of vaccine against COVID-19 using enzyme immunoassay using the Sunrise Tecan microplate photometer (Austria). The material is participants' plasma, obtained by the standard method. Blood sampling performed 4 times: immediately before the first dose of vaccine, on day 42, 90 days and 180 days after booster dose of vaccine. Booster dose of vaccine against coronavirus infection performing using approved and licensed vaccine Soberana Plus (Republic of Cuba). Venous blood sampling performing standardly. All study participants are informed about the study objectives and upcoming procedures, and all of them given informed written consent to participate the study.

A reagent kit manufactured by Vector-Best (Russian Federation) and designed for enzyme immunoassay for quantitative detection of SARS-CoV-2 class G immunoglobulins, SARS-CoV-2-IgG quantitative ELISA-BEST, D-5505 SARS-CoV-2-IgG (series 5, 6) РУ № РЗН 2022/17065Т used for immunoassay. The "SARS-CoV-2-IgG quantitative ELISA-BEST" reagent kit design uses recombinant full-length trimerized S glycoprotein (Spike) of the SARS-CoV-2 virus derived from a eukaryotic expression system. The protein molecule+ consists of two subunits, S1 containing the RBD domain and S2. The reagent kit "SARS-CoV-2-IgG quantitative ELISA-BEST" detects the pool of immunoglobulin class G synthesized to all antigenic determinants of protein S including the RBD-domain.

The quantification of the SARS-CoV-2 antibody assay is based on the WHO First International Standard (NIBSC code:20/136) and expressed in international units (BAU/ml).

Analytical characteristics of reagent kit "SARS-CoV-2-IgG quantitative ELISA-BEST (series 5, 6)" were: Linearity - within 90-110%, considering the analytical results at wavelengths 405 nm and 415 nm - within the concentration range IgG к SARS-CoV-2 10-5000 BAU/ml; Reproducibility: the coefficient of variation does not exceed 8%). The "opening" test - within 90-110% (samples with absorbances lower than 90% of the cut-off value are considered negative and samples with absorbances higher than 110% of the cut-off value are considered positive. The samples with absorbance in the range of 90-110% of cut-off value are equivocal). Analytical sensitivity - minimal detectable concentration of IgG to SARS-CoV-2 does not exceed 1.0 BAU/ml.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 y.o.;
2. More that 4 months after the previous vaccination against COVID-19;
3. No COVID-19 infection registered within 30 days prior to Soberana Plus administration.

Exclusion Criteria:

1. Age less than 18 y.o. or more than 80 y.o.;
2. Less than 4 months after the previous vaccination against COVID-19;
3. COVID-19 infection registered within 30 days prior to Soberana Plus administration.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-12-09 (Actual); Primary Completion 2023-03-10 (Estimated); Study Completion 2023-07-28 (Estimated)

PRIMARY OUTCOMES:
IgG level assessment | 42 days after booster dose administration
  The quantification of the SARS-CoV-2 antibody assay
IgG level assessment | 90 days after booster dose administration
  The quantification of the SARS-CoV-2 antibody assay
IgG level assessment | 180 days after booster dose administration
  The quantification of the SARS-CoV-2 antibody assay

CONTACTS AND LOCATIONS:
Overall Officials: Igor Stoma, MD, Study Chair — Gomel state medical university, Gomel, Province, Belarus, 246000; Olga Osipkina, Principal Investigator — Gomel State Medical University, Gomel, Province, Belarus, 246000
Locations (1):
- Gomel State Medical University, Homyel, Belarus

IPD SHARING:
Plan to Share IPD: No